CLINICAL TRIAL: NCT01815710
Title: Best Strategies for Implementation of Clinical Pathways in Emergency Department Settings
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Mona Jabbour, Vice-Chief/Chair, Department of Pediatrics, Children's Hospital of Eastern Ontario
Other Study IDs: DCO150GP
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Asthma; Diarrhea & Vomiting
Keywords: Clinical Pathways; Knowledge translation; Evaluation
MeSH Terms: conditions — Asthma; Diarrhea; Vomiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vomiting & Diarrhea: Alberta Health Services Acute Childhood Vomiting & Diarrhea Pathway
  Interventions: Other: Vomiting & Diarrhea Pathway
- Pediatric Asthma Clinical Pathway: Pediatric Asthma Clinical Pathway
  Interventions: Other: Pediatric Asthma Clinical Pathway

INTERVENTIONS:
Other: Pediatric Asthma Clinical Pathway — Implementation of a clinical pathway outlining standardized, evidence-based care for pediatric patients with asthma. These clinical pathways use organized, time-sequenced interventions to achieve optimal patient outcomes.
  Groups: Pediatric Asthma Clinical Pathway
Other: Vomiting & Diarrhea Pathway — Implementation of a clinical pathway outlining standardized, evidence-based care for pediatric patients with vomiting and diarrhea. These clinical pathways use organized, time-sequenced interventions to achieve optimal patient outcomes.
  Groups: Vomiting & Diarrhea

SUMMARY:
An Ontario-wide study to identify best strategies to promote uptake of high quality, expert developed Clinical Pathways (CPs) within Emergency Departments.

The investigators will work with 16 Community EDs across Ontario to i) tailor an implementation strategy that works for each ED, ii) assist with the implementation of one pediatric emergency CP (Asthma or Gastroenteritis) at each site, and iii) evaluate the impact on health professionals, patient outcomes and economic costs. The investigators will conduct a 3.5 - year mixed methods health services research project with four study objectives: 1) to design a theory-based and knowledge user-informed intervention strategy to successfully implement two provincial pediatric emergency clinical pathways into practice in community Emergency Departments (EDs); 2) to evaluate the effectiveness of this implementation strategy; 3) to conduct a process evaluation to assess the implementation strategy; and 4) to conduct an economic analysis to evaluate implementation costs and benefits.

DETAILED DESCRIPTION:
To meet the first objective, we will use Michie's Theoretical Domains Framework (TDF) to identify and organize CP-relevant behaviours. We will conduct qualitative interviews, guided by the TDF and involving knowledge users from participating sites, to identify barriers and facilitators for change relevant to the proposed CP implementation. Experience from other implementation initiatives will also be used to guide the intervention. An intervention mapping technique will be used to select and organize appropriate strategies to affect behaviour changes. Further input will be sought from knowledge user site partners. The intervention will begin with a site visit to assess readiness for adoption, infrastructure requirements, and ability to implement the pathway.

To meet objective two, we will use a cluster randomized control trial (RCT) design, through measurement of relevant clinical and process outcomes in 16 community EDs in Ontario. Using a balanced incomplete block design, we will study this implementation intervention with two clinical pathways: i) Asthma and ii) Vomiting & Diarrhea (V&D). We will recruit and randomize 16 community EDs to receive the intervention for one of the CPs and serve as control for the alternate pathway. Primary clinical outcomes for each CP include the following: i) Asthma: the proportion of asthmatic patients with moderate to severe exacerbation who received steroids within 60 minutes from ED presentation; and ii) V&D: the proportion of children with mild to moderate dehydration treated with oral rehydration therapy. The primary process outcome measure will be the presence of an appropriately completed CP, as per pre-defined criteria, on the chart for relevant patients. Secondary clinical outcomes include disease-specific treatments, ED length of stay, revisits and hospitalizations. Secondary process outcomes include CP use based on shift-level data relating to the busyness of the ED. A mixed methods evaluation will be used to assess clinical and process outcomes. Data sources include chart audits, administrative databases, environmental scans and knowledge user interviews. Sample size calculations for the primary process outcome yielded the highest number of required charts. A total sample size of 6400 patient charts is required to detect an absolute difference of 12% between control and intervention hospitals using a two-sided test at the 5% level of significance.

To meet objective three, a process log will be used to track progress with site deadline targets, implementation issues, degree of uptake, local adaptations and adherence.

And finally, to meet objective four, comparisons of CP implementation and health care costs will be done for all patients with Asthma or V&D in the pre and post implementation phases at all sites. Additional costs and outcomes will be synthesized in an incremental cost-effectiveness ratio (ICER) comparing intervention and control sites. Cost-effectiveness analyses (CEAs) will be done to relate ICERs to the primary clinical outcome for each CP.

ELIGIBILITY:
Inclusion Criteria:

* Selecting from 149 community EDs in Ontario, we will recruit EDs that do not have a CP in place for either Pediatric Asthma or Pediatric V&D. To minimize contamination between sites, we will request data from Health Force Ontario, an organization that assists with physician coverage at different EDs, to ensure ED physicians are not working at more than one study site. An additional inclusion criterion is commitment to the implementation intervention by an administrative lead on behalf of the hospital. Specific inclusion/exclusion criteria for use with patients have been defined for each CP.
* Medical records departments at each site will be asked to pull relevant charts, using International Statistical Classification of Diseases and Related Health Problems (ICD)-10 codes for all diagnoses related to our index conditions (Asthma and with V&D) during the defined study periods. In our experience, this approach has worked successfully with community ED studies. Chart auditors will review all records to ensure eligibility criteria are met. All retrieved and eligible patient charts will be audited.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community hospitals in a variety of local health integration networks across Ontario (very high to low volume).
Sampling Method: Non-Probability Sample
Enrollment: 6330 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Received appropriate care based on evidence-based treatments recommended in the CP. | 18 months
  The proportion of pediatric patients with asthma and V&D who received appropriate care based on evidence-based treatments recommended in the CP.

SECONDARY OUTCOMES:
Asthma - PRAM | 18 months
  Asthma CP intervention will include: 1) documentation of a Pre-school Respiratory Assessment Measure (PRAM) score.
V&D - Gorelick and intravenous therapy. | 18 months
  For the V&D CP intervention, secondary clinical outcomes will include: 1) documentation of a Gorelick score for dehydration; and 2) the proportion of children treated with intravenous therapy for rehydration.

OTHER OUTCOMES:
Completed CP on relevant patient charts. | 18 months
  Our primary process outcome will be a completed CP on relevant patient charts. Each CP will be reviewed to determine required clinical care elements to achieve the CP goals, and completion criteria will be defined to guide determination of one of three grades: 1) initial, with the CP started with little or no documentation; 2) partial, with some but incomplete documentation; or 3) full, meeting sufficient requirements for CP success. Because the busyness of a given shift may affect CP use decisions, a secondary outcome will be CP use for relevant patients, adjusted for shift-level ED data.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Jabbour, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jabbour M, Newton AS, Johnson D, Curran JA. Defining barriers and enablers for clinical pathway implementation in complex clinical settings. Implement Sci. 2018 Nov 12;13(1):139. doi: 10.1186/s13012-018-0832-8. PMID 30419942
- [Derived] Jabbour M, Curran J, Scott SD, Guttman A, Rotter T, Ducharme FM, Lougheed MD, McNaughton-Filion ML, Newton A, Shafir M, Paprica A, Klassen T, Taljaard M, Grimshaw J, Johnson DW. Best strategies to implement clinical pathways in an emergency department setting: study protocol for a cluster randomized controlled trial. Implement Sci. 2013 May 22;8:55. doi: 10.1186/1748-5908-8-55. PMID 23692634